CLINICAL TRIAL: NCT00300248
Title: The Improving Care of Acute Lung Injury Patients (ICAP) Study
Brief Title: Long-Term Results in Mechanically Ventilated Individuals With Acute Lung Injury/Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dale Needham, Professor, Johns Hopkins University
Other Study IDs: 1329; P50HL073994-03 (NIH); R01HL088045 (NIH)
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Failure; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute lung injury/acute respiratory distress syndrome (ALI/ARDS) is a severe lung condition that causes respiratory failure. Individuals with ALI/ARDS often require the use of a respirator or artificial breathing machine, known as a mechanical ventilator, while in an intensive care unit (ICU). Past research has shown that improved short-term clinical outcomes result from the use of a protective mechanical ventilation technique for the lungs. This study will evaluate the effects of lower tidal volume ventilation, and other aspects of critical illness and ICU care, on the long-term clinical outcomes of individuals with ALI/ARDS.

DETAILED DESCRIPTION:
ALI/ARDS is a life-threatening condition that involves inflammation of the lungs and fluid accumulation in the air sacs, which leads to low blood oxygen levels and respiratory failure. Common causes include pneumonia, septic shock, and lung trauma. Symptoms usually develop within 24 to 48 hours of the original injury or illness, and most patients require immediate care in an intensive care unit (ICU). The main form of treatment for ALI/ARDS is the delivery of oxygen and a continuous level of pressure to the damaged lungs through mechanical ventilation. Past research has shown that lower tidal volume ventilation (LTVV), a protective ventilator management technique in which lower volumes of oxygen are administered, improves short-term clinical outcomes in individuals with ALI/ARDS. However, the long-term impact of LTVV remains unknown. The purpose of this study is to evaluate the effects of LTVV on long-term outcomes in individuals with ALI/ARDS.

This study will enroll individuals admitted to an ICU who have been recently diagnosed with ALI/ARDS. Once enrolled, participants' medical records will be reviewed for demographic and medical information. Participants will be examined to determine level of cognition and delirium. Questionnaires will be used to assess the participant's status prior to ICU admittance, including level of hearing, physical functioning, quality of life, employment, and living status. Questionnaires will be given to participants as well as a close contact to increase the reliability of feedback. While in the ICU, participants will receive normal clinical care. Data on laboratory tests, mechanical ventilator settings, arterial blood gas values, and medical status will be collected throughout the ICU stay. Information regarding the medical staff-to-patient ratio and the use of different medical treatments and therapies will also be collected by reviewing medical records and interviewing nurses. Follow-up evaluations, lasting approximately four hours each, will occur 3, 6, 12, 24, 36, 48 and 60 months following the ALI/ARDS diagnosis. At each follow-up visit, participants will undergo a physical examination, and standardized surveys and tests will be used to assess medical outcomes, organ impairment, pulmonary function, mental function, and quality of life. If participants are unable to return to the research clinic for the follow-up evaluations, visits may occur at their home or over the phone.

The original 2-year follow-up duration, for which participants were consented, was subsequently extended to allow 5-year follow-up. In recruiting these previously consented participants into the 5-year follow-up extension, they will be randomized to selected recruitment strategies (e.g., different mailing and telephone strategies) in order to gain insight regarding the most effective methods of recruiting participants.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the ICU
* Receiving mechanical ventilation
* Meets criteria for the diagnosis of ALI/ARDS, as defined by the American-European Consensus Conference

Exclusion Criteria:

* Received diagnosis of ALI/ARDS more than 96 hours prior to study entry
* Received more than five days of mechanical ventilation during the present hospitalization prior to study entry
* Pre-existing ALI/ARDS for more than 24 hours when transferred to the study ICU
* Pre-existing illness with a life expectancy of less than six months
* Any limitations in ICU care at study entry (e.g., no vasopressor)
* Previous lung resection
* Inability to speak or understand English
* No fixed address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 13 critical care units at 4 academic hospitals in Baltimore, MD
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2004-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mortality | Measured at Months 3, 6, 12, 24, 36, 48 and 60

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Pronovost, MD, PhD, Principal Investigator — Johns Hopkins University; Dale M. Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Bayview Medical Center, Baltimore, Maryland

REFERENCES:
- [Background] Needham DM, Dennison CR, Dowdy DW, Mendez-Tellez PA, Ciesla N, Desai SV, Sevransky J, Shanholtz C, Scharfstein D, Herridge MS, Pronovost PJ. Study protocol: The Improving Care of Acute Lung Injury Patients (ICAP) study. Crit Care. 2006 Feb;10(1):R9. doi: 10.1186/cc3948. PMID 16420652
- [Background] Fan E, Needham DM, Stewart TE. Ventilatory management of acute lung injury and acute respiratory distress syndrome. JAMA. 2005 Dec 14;294(22):2889-96. doi: 10.1001/jama.294.22.2889. PMID 16352797
- [Background] Needham DM, Dowdy DW, Mendez-Tellez PA, Herridge MS, Pronovost PJ. Studying outcomes of intensive care unit survivors: measuring exposures and outcomes. Intensive Care Med. 2005 Sep;31(9):1153-60. doi: 10.1007/s00134-005-2656-7. Epub 2005 May 21. PMID 15909169
- [Background] Dowdy DW, Needham DM, Mendez-Tellez PA, Herridge MS, Pronovost PJ. Studying outcomes of intensive care unit survivors: the role of the cohort study. Intensive Care Med. 2005 Jul;31(7):914-21. doi: 10.1007/s00134-005-2657-6. Epub 2005 May 21. PMID 15909168
- [Background] Dowdy DW, Eid MP, Sedrakyan A, Mendez-Tellez PA, Pronovost PJ, Herridge MS, Needham DM. Quality of life in adult survivors of critical illness: a systematic review of the literature. Intensive Care Med. 2005 May;31(5):611-20. doi: 10.1007/s00134-005-2592-6. Epub 2005 Apr 1. PMID 15803303
- [Background] Dowdy DW, Eid MP, Dennison CR, Mendez-Tellez PA, Herridge MS, Guallar E, Pronovost PJ, Needham DM. Quality of life after acute respiratory distress syndrome: a meta-analysis. Intensive Care Med. 2006 Aug;32(8):1115-24. doi: 10.1007/s00134-006-0217-3. Epub 2006 Jun 17. PMID 16783553
- [Background] Desai SV, Boucher K, Fan E, Needham DM. Long-term outcomes after acute lung injury. Contemporary Critical Care. 2006;4:1-10
- [Background] Moss RE. Affordable health care. Crit Care Med. 2004 Dec;32(12):2564; author reply 2564. doi: 10.1097/01.ccm.0000153900.88044.b5. No abstract available. PMID 15599184
- [Background] Ciesla N, Barbe C, Patel N, Mendez-Tellez PA, Dennison CR, Needham DM. Physical therapy for the intensive care unit: implications based on evaluation of critical care management of 150 acute lung injury/acute respiratory distress syndrome patients. Cardiopulmonary Physical Therapy Journal 17(4): 142, 2006.
- [Background] Needham DM, Wang W, Desai SV, Mendez-Tellez PA, Dennison CR, Sevransky J, Shanholtz C, Ciesla N, Spillman K, Pronovost PJ. Intensive care unit exposures for long-term outcomes research: development and description of exposures for 150 patients with acute lung injury. J Crit Care. 2007 Dec;22(4):275-84. doi: 10.1016/j.jcrc.2007.02.001. Epub 2007 Jun 27. PMID 18086397
- [Background] Dennison CR, Mendez-Tellez PA, Wang W, Pronovost PJ, Needham DM. Barriers to low tidal volume ventilation in acute respiratory distress syndrome: survey development, validation, and results. Crit Care Med. 2007 Dec;35(12):2747-54. doi: 10.1097/01.CCM.0000287591.09487.70. PMID 17901838
- [Background] Fan E, Shahid S, Kondreddi VP, Bienvenu OJ, Mendez-Tellez PA, Pronovost PJ, Needham DM. Informed consent in the critically ill: a two-step approach incorporating delirium screening. Crit Care Med. 2008 Jan;36(1):94-9. doi: 10.1097/01.CCM.0000295308.29870.4F. PMID 18090168
- [Background] Umoh NJ, Fan E, Mendez-Tellez PA, Sevransky JE, Dennison CR, Shanholtz C, Pronovost PJ, Needham DM. Patient and intensive care unit organizational factors associated with low tidal volume ventilation in acute lung injury. Crit Care Med. 2008 May;36(5):1463-8. doi: 10.1097/CCM.0b013e31816fc3d0. PMID 18434907
- [Background] Dowdy DW, Dinglas V, Mendez-Tellez PA, Bienvenu OJ, Sevransky J, Dennison CR, Shanholtz C, Needham DM. Intensive care unit hypoglycemia predicts depression during early recovery from acute lung injury. Crit Care Med. 2008 Oct;36(10):2726-33. doi: 10.1097/CCM.0b013e31818781f5. PMID 18766087
- [Background] Fan E, Khatri P, Mendez-Tellez PA, Shanholtz C, Needham DM. Review of a large clinical series: sedation and analgesia usage with airway pressure release and assist-control ventilation for acute lung injury. J Intensive Care Med. 2008 Nov-Dec;23(6):376-83. doi: 10.1177/0885066608324293. Epub 2008 Sep 19. PMID 18805857
- [Background] Sevransky JE, Martin GS, Mendez-Tellez P, Shanholtz C, Brower R, Pronovost PJ, Needham DM. Pulmonary vs nonpulmonary sepsis and mortality in acute lung injury. Chest. 2008 Sep;134(3):534-538. doi: 10.1378/chest.08-0309. Epub 2008 Jul 18. PMID 18641112
- [Result] Dowdy DW, Bienvenu OJ, Dinglas VD, Mendez-Tellez PA, Sevransky J, Shanholtz C, Needham DM. Are intensive care factors associated with depressive symptoms 6 months after acute lung injury? Crit Care Med. 2009 May;37(5):1702-7. doi: 10.1097/CCM.0b013e31819fea55. PMID 19357507
- [Result] Murphy DJ, Howard D, Muriithi A, Mendez-Tellez P, Sevransky J, Shanholtz C, Netzer G, Pronovost PJ, Needham DM. Red blood cell transfusion practices in acute lung injury: what do patient factors contribute? Crit Care Med. 2009 Jun;37(6):1935-40. doi: 10.1097/CCM.0b013e3181a0022d. PMID 19384204
- [Derived] Kamdar BB, Sepulveda KA, Chong A, Lord RK, Dinglas VD, Mendez-Tellez PA, Shanholtz C, Colantuoni E, von Wachter TM, Pronovost PJ, Needham DM. Return to work and lost earnings after acute respiratory distress syndrome: a 5-year prospective, longitudinal study of long-term survivors. Thorax. 2018 Feb;73(2):125-133. doi: 10.1136/thoraxjnl-2017-210217. Epub 2017 Sep 16. PMID 28918401
- [Derived] Needham DM, Yang T, Dinglas VD, Mendez-Tellez PA, Shanholtz C, Sevransky JE, Brower RG, Pronovost PJ, Colantuoni E. Timing of low tidal volume ventilation and intensive care unit mortality in acute respiratory distress syndrome. A prospective cohort study. Am J Respir Crit Care Med. 2015 Jan 15;191(2):177-85. doi: 10.1164/rccm.201409-1598OC. PMID 25478681
- [Derived] Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ. Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ. 2012 Apr 5;344:e2124. doi: 10.1136/bmj.e2124. PMID 22491953